CLINICAL TRIAL: NCT00260520
Title: Low Molecular Weight Heparin Vs No Treatment in Pregnant Women With Previous Preeclampsia or Fetal Growth Restriction Who Were Heterozygote for Factor V Leiden or Prothrombin Gene G20210A Mutation
Brief Title: LMWH to Prevent Preeclampsia and Fetal Growth Restriction
Status: Terminated | Type: Observational
Sponsor: University of Florence (Other)
Other Study IDs: 06-03-1942
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2006-03-06 (Estimated); Status verified 2003-12

CONDITIONS: Preeclampsia
Keywords: Low molecular weight heparin; Preeclampsia; Fetal Growth Restriction; Thrombophilia; Factor V Leiden; G20210A prothrombin gene mutation
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Thrombophilia | interventions — Dalteparin

INTERVENTIONS:
Drug: Dalteparin

SUMMARY:
The objective of this trial will be to determine whether prophylactic low-molecular weight heparin therapy in pregnant women with the heterozygous Factor V Leiden and G20210A prothrombin gene mutations thrombophilia and a history of severe preeclampsia and/or severe fetal growth restriction reduces the risk of the composite outcome of preeclampsia, fetal growth restriction, or both.

DETAILED DESCRIPTION:
The objective of this trial will be to determine whether prophylactic low-molecular weight heparin therapy in pregnant women with the heterozygous Factor V Leiden and G20210A prothrombin gene mutations thrombophilia and a history of severe preeclampsia and/or severe fetal growth restriction reduces the risk of the composite outcome of preeclampsia, fetal growth restriction, or both. We also will assess the effect of treatment on other indicators of maternal and neonatal complications, and the growth of fetal body composition in terms of fat and lean body mass.

ELIGIBILITY:
Inclusion Criteria:

* Previous severe preeclampsia
* Previous severe fetal growth restriction
* Heterozygous Factor V Leiden
* Heterozygous G20210A prothrombin gene mutations

Exclusion Criteria:

* renal disease
* chronic hypertension
* preexisting diabetes mellitus
* homozygosity for Factor V Leiden
* homozygosity for prothrombin G20210A mutation
* hyperhomocysteinemia
* protein C deficency
* protein S deficency
* antithrombin deficiency
* positive anticardiolipin antibodies
* positive lupus anticoagulant

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2002-01; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Mello, MD, Study Director — Department of Gynecology, Perinatology and Human Reproduction, University of Florence, Italy